CLINICAL TRIAL: NCT01107353
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Imipramine Pamoate Capsules, 75 mg, Under Fasted Conditions
Brief Title: Bioequivalency Study of Imipramine Pamoate 75 mg Capsules Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IMIP-C75-PVFS-1
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Imipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Imipramine Pamoate, then Tofranil-PM (Active Comparator): First 75 mg imipramine pamoate capsule, then 75 mg Tofranil-PM capsule (after washout period)
  Interventions: Drug: Imipramine Pamoate
- First Tofranil PM, then imipramine pamoate (Active Comparator): First 75 mg Tofranil-PM capsule, then 75 mg imipramine pamoate capsule (after washout period)
  Interventions: Drug: Imipramine Pamoate

INTERVENTIONS:
Drug: Imipramine Pamoate — 75 mg capsule
  Other Names: TOFRANIL-PM

SUMMARY:
The objective of this study was to prove the bioequivalence of Imipramine Pamoate 75 mg Capsules under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to imipramine pamoate or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | First Imipramine Pamoate, Then Tofranil-PM | First Tofranil PM, Then Imipramine Pamoate
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Positive Drug Screen | 1 | 0

BASELINE CHARACTERISTICS:
Population: Normal healthy volunteers
Groups:
- Total: Total of all reporting groups
Arm/Group | First Imipramine Pamoate, Then Tofranil-PM | First Tofranil PM, Then Imipramine Pamoate | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.41 (7.65) | 28.41 (7.65) | 28.41 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 17 | 36
  White | 0 | 3 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence Determined by Statistical Comparison Cmax
Description: Blood samples were collected pre-dose and at intervals over 120 hours after each dose
Time Frame: 33 Days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | First Imipramine Pamoate, Then Tofranil-PM | First Tofranil PM, Then Imipramine Pamoate
Number analyzed (Participants) | 19 | 19
ng/mL | 11.5 (7.48) | 11.3 (7.03)

ADVERSE EVENTS:
Time Frame: 33 days
Arm/Group | First Imipramine Pamoate, Then Tofranil-PM | First Tofranil PM, Then Imipramine Pamoate
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days